CLINICAL TRIAL: NCT03147339
Title: The Effects of Restricted Dietary of Advanced Glycation End Products(AGEs) on the Glycemic Control, Oxidative Stress and Systemic-inflammation in Patients With Metabolic.
Brief Title: The Effects of Restricted Dietary of AGEs on the Glycemic Control, Oxidative Stress and Inflammation
Acronym: AGEs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Azita Hekmatdoost (Other)
Responsible Party: Sponsor-Investigator, Dr Azita Hekmatdoost, Principal Investigator, National Nutrition and Food Technology Institute
Organization: National Nutrition and Food Technology Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NNFTRI691
Record Dates: First submitted 2017-04-30; First posted 2017-05-10 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Metabolic Syndrome
Keywords: AGEs( Advanced glycation end products)
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AGEs restricted diet (Experimental): Low calorie diet + AGEs restricted diet
  Interventions: Other: AGEs restricted diet
- control (No Intervention): Low calorie diet

INTERVENTIONS:
Other: AGEs restricted diet — Diet modification to reduce advanced glycation end products in diet. for example to change ways of cooking, time of cooking and also omit some foods.
  Arms: AGEs restricted diet

SUMMARY:
To evaluate the effects of dietary restriction of advanced glycated end products (AGEs) on glycemic control, oxidative stress and systemic inflammation, in a randomized, 44 subjects with metabolic syndrome for 8 weeks.Both groups will be advised to follow same low energy diet and no changing in physical activity pattern.Parameters related to metabolic syndrome, anthropocentric factors, oxidative stress(Malondialdehyde), CML(AGEs factor in blood) and systemic inflammation factors (hs-CRP وTNF-α ) will be measured at the baseline and at the end of the study.

DETAILED DESCRIPTION:
Metabolic syndrome (MS) is a cluster of cardiovascular risk factor abnormalities associated with increased risk of type 2 diabetes mellitus, cardiovascular disease, and all-cause mortality. Non-enzymatic glycation plays an important role in the development of physiological and pathophysiological processes such as aging, diabetes, atherosclerosis, and chronic renal failure. Preventing glycation can minimize diabetic complications. Advanced glycation end products (AGEs) are formed endogenously when the carbonyl groups of reducing sugars nonenzymatically react with the free amino groups on proteins. AGEs are generated in vivo as a normal consequence of metabolism, but their formation is accelerated under conditions of hyperglycemia, hyperlipidemia and increased oxidative stress. It can also form in food processing and the variety and the amount of dietary AGEs (dAGE) depend on food nutrients, the heating used in food processing, pH conditions, presence of some metal ions (Cu++, Fe++) and water content. In this study 2 groups of metabolic syndrome patients(22 in each group) will receive same low calorie diet and one of the groups plus restricted dietary AGEs according to the international references.Along 8 weeks the investigators will talk to each patient by phone and every months the participants will come and the investigators will take anthropocentric measurements and the recommendations for diets will review. The three-day 24-hour recall food questionnaire will take at first,middle and the end of program.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age
* having three of the following five features: Increased waist circumference (≥102 cm in men and ≥88 cm in women), elevated TG (≥150 mg/dl), reduced HDL-C (≤40 mg/dl in men and ≤50 mg/dl in women), elevated blood pressure (≥130/85 mm Hg or on treatment for hypertension) and elevated glucose (≥100 mg/dl), according to the National Cholesterol Education Program Adult Treatment Panel III report

Exclusion Criteria:

* history of allergy
* clinically diagnosed renal, pituitary, thyroid, infections and inflammations, cancer and using of insulin, using multivitamin mineral and vitamin B6 suplements.
* Using any
* history of cancers.
* pregnancy, lactation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Serum Levels of carboxymethyl-lysine(CML) | 8 weeks
  specific serum AGEs

CONTACTS AND LOCATIONS:
Overall Officials: National Nutrition and Food Technology Research Institute, Study Director — Shahid Beheshti University of Medical Sciences
Locations (1):
- National Nutrition and Food Technology Research Institute, Tehrān, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: No